CLINICAL TRIAL: NCT03337906
Title: A Descriptive and Observational Study of Long-term Outcomes of HIV-1 Infection in Persons Who Become HIV-1 Infected After Enrollment in HIV-1 Vaccine Trials
Brief Title: An Observational Study of Long-term Outcomes of HIV-1 Infection in Persons Who Become HIV-1 Infected After Enrollment in HIV-1 Vaccine Trials
Status: Completed | Type: Observational
Sponsor: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Other Study IDs: HVTN 802
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants infected with HIV-1: Persons who become HIV-1 infected after enrollment in HIV-1 vaccine trials
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
An observational study of long-term outcomes of HIV-1 infection in persons who become infected after enrollment in HIV-1 vaccine trials

DETAILED DESCRIPTION:
A descriptive and observational study of long-term outcomes of HIV-1 infection in persons who become HIV-1 infected after enrollment in HIV-1 vaccine trials

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria in order to be eligible for inclusion in the study:

  1. Confirmation of HIV-1 infection after enrollment in an HVTN vaccine trial in which HIV-1 infection constituted an endpoint, according to the diagnostic algorithm specified in the parent protocol.
  2. Ability and willingness to provide written informed consent to participate in the study.
  3. Ability and willingness to adhere to the on-study follow-up schedule.
  4. Ability and willingness to provide adequate information for locator purposes.
  5. Participants who are currently on ART or who previously received antiretrovirals as part of post-exposure prophylaxis, pre-exposure prophylaxis, or previous treatment regimen will be eligible for inclusion in this protocol. Their previous treatment history will be collected. If a participant has been on ART for more than 2 years, please consult with the protocol team leadership prior to enrollment.
  6. For participants initiating ART, agreement of participant and PHCP to initiate potent and durable ART regimens in accordance with local and international guidelines. Examples of potent and durable regimens are provided in Appendix H. Participants who initiate ART not consistent with regimens outlined in Appendix H may enroll with permission of the protocol chair or designee(s).

     Exclusion Criteria:
* Persons who meet the following criteria will be excluded from the study:

  1. Any medical, psychiatric, alcohol/drug dependency or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence or a participant's ability to give informed consent.
  2. Participants who meet these additional criteria will be excluded from the study:
* Participants undergoing acute therapy for serious medical illnesses (in the opinion of the site investigator) within 14 days prior to initiation of ART.
* Participants with chronic, acute, or recurrent infections that are serious (in the opinion of the site investigator).
* Participants who must continue with chronic (maintenance) therapy (e.g., tuberculosis [TB], pneumocystis pneumonia [PCP]), must have completed at least 14 days of therapy and be clinically stable prior to initiation of ART.
* Oral and vaginal candidiasis, mucocutaneous herpes simplex, and other minor illnesses, as defined by the site investigator, present no restriction to eligibility.
* Participants undergoing radiation therapy, systemic chemotherapy, or receiving an immunomodulator within 45 days prior to initiation of ART. (A tapering course of corticosteroids as acute therapy for PCP or other conditions is an exception.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both vaccine and placebo recipients in HVTN trials in which HIV infection constitutes an endpoint (eg, test-of-concept, phase 2 and 3) who become HIV-1 infected after enrollment in the parent study and who meet the inclusion criteria may be offered enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2008-07-11 (Actual); Primary Completion 2015-07-11 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Measure plasma HIV-1 RNA levels and CD4+ T cell counts longitudinally | 8 years
  Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.
Measure time to initiation of ART | 8 years
  Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.
Measure time to HIV-1 related clinical events | 8 years
  Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.
  Responses from ELISpot assays will be reported as the number of spot-forming cells Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.
Proportion of individuals with plasma HIV-1 RNA level <50 copies/mL at 24 weeks after initiation of ART | 8 years
  Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.
  Responses from ELISpot assays will be reported as the number of spot-forming cells Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.

SECONDARY OUTCOMES:
Time from initiation of ART to treatment failure due to virologic, immunologic, and clinical reasons | 8 years
  Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.
Occurrence of HIV/AIDS associated events, including death | 8 years
  Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.
Proportion of subjects with HIV-1 RNA level <50 copies/mL post-initiation of ART; log change in plasma HIV-1 RNA levels and change in CD4+ T cell levels between baseline (at initiation of ART) and post-initiation of ART | 24, 48, 96, and 144 weeks
  Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.
Adherence information collected at 24, 48, 96, and 144 weeks following initiation of ART | 24, 48, 96, and 144 weeks
  Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.
Side effects collected at 24, 48, 96, and 144 weeks following initiation of ART | 24, 48, 96, and 144 weeks
  Blood samples will be processed for PBMCs and then cryopreserved. These specimens will be stimulated with synthetic HIV-1 peptide pools. This process will allow ex vivo HIV-specific T-cell responses to be assessed by IFN-γ ELISpot and/or flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Sobieszcyk, Study Chair — Columbia University
Locations (21):
- United States (13):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - UIC Project WISH CRS, Chicago, Illinois
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health Clinical Research Site CRS, Boston, Massachusetts
  - NY Blood Ctr./Union Square CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - NY Blood Ctr./Bronx CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, New York, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- Unidad de Vacunas IDCP-COIN-DIGECITSS CRS, Santo Domingo, Dominican Republic
- Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince, Haiti
- ACSA CRS, Iquitos, Maynas, Peru
- Maternal-Infant Studies Center (CEMI) CRS, San Juan, Puerto Rico
- South Africa (4):
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - eThekwini CRS, Durban, KwaZulu-Natal
  - Aurum Institute Klerksdorp CRS, Klerksdorp, North West
  - Emavundleni CRS, Cape Town, Western Cape